CLINICAL TRIAL: NCT01846962
Title: COMPARISON OF TREATMENT FOR PEDIATRIC EOSINOPHILIC ESOPHAGITIS: A RANDOMIZED CLINICAL TRIAL (DIETETIC Versus TOPICAL STEROIDS)
Brief Title: Dietetic Versus Topical Steroids for Pediatric Eosinophilic Esophagitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Salvatore Oliva, MD, Azienda Policlinico Umberto I
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pediatric-EoE
Record Dates: First submitted 2013-04-30; First posted 2013-05-06 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic esophagitis (EoE); budesonide; fluticasione; six-foods elimination diet
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Budesonide; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- six-foods elimination diet (Experimental): six-foods elimination diet. The standard panel of foods tested included the 6 most common allergenic foods in childhood (cow's milk, egg, soy, wheat, peanuts, fish), plus foods that were suspiciously implicated in triggering an allergic reaction referred by patients or their parents. Both perennial (dust mite, Parietaria, Alternaria, cat and dog dander) and seasonal (grass pollen including Graminaceae, Olea europea, Platanus) aeroallergens have been tested.
  Interventions: Behavioral: six-foods elimination diet
- fluticasone (Experimental): The administered dose of topical steroid was 440mcg or 880mcg/day (<150 cm or >150 cm). Patients were trained to swallow puffs and to non eat or drink fo 30 minutes after ingestion. Patients noncompliant with therapy, monthly assessed by Pediatric Allergologists, were withdrawn from the study.
  Interventions: Drug: Fluticasone
- Budesonide (Experimental): The administered dose of topical steroid was 400mcg/day or 800 mcg/day (<150 cm or >150 cm). Patients were trained to swallow puffs and to non eat or drink fo 30 minutes after ingestion. Patients noncompliant with therapy, monthly assessed by Pediatric Allergologists, were withdrawn from the study.
  Interventions: Drug: Budesonide
- Oral Viscous Budesonide (OVB) (Experimental): The administered dose of topical steroid was 1 or mg/day (<150 cm or >150 cm). Patients were trained to prepare a homemade suspension of OVB prepared by mixing inhaled budesonide with viscous solutions of sodium alginate and to non eat or drink fo 30 minutes after ingestion. Patients noncompliant with therapy, monthly assessed by Pediatric Allergologists, were withdrawn from the study.
  Interventions: Drug: Oral Viscous Budesonide (OVB)

INTERVENTIONS:
Drug: Budesonide — The administered dose of topical steroid was 400mcg or 800mcg/day (<150 cm or >150 cm). Patients were trained to swallow puffs and to non eat or drink fo 30 minutes after ingestion. Patients noncompliant with therapy, monthly assessed by Pediatric Allergologists, were withdrawn from the study.
  Arms: Budesonide
Drug: Fluticasone — The administered dose of topical steroid was 440mcg or 880mcg/day (<150 cm or >150 cm). Patients were trained to swallow puffs and to non eat or drink fo 30 minutes after ingestion. Patients noncompliant with therapy, monthly assessed by Pediatric Allergologists, were withdrawn from the study.
  Arms: fluticasone
Behavioral: six-foods elimination diet — six-foods elimination diet. The standard panel of foods tested included the 6 most common allergenic foods in childhood (cow's milk, egg, soy, wheat, peanuts, fish), plus foods that were suspiciously implicated in triggering an allergic reaction referred by patients or their parents. Both perennial (dust mite, Parietaria, Alternaria, cat and dog dander) and seasonal (grass pollen including Graminaceae, Olea europea, Platanus) aeroallergens have been tested.
  Arms: six-foods elimination diet
Drug: Oral Viscous Budesonide (OVB) — The administered dose of topical steroid was 1mg/day or 2mg/day (<150 cm or >150 cm). Patients were trained to prepare a homemade suspension of OVB prepared by mixing inhaled budesonide with viscous solutions of sodium alginate and to non eat or drink fo 30 minutes after ingestion. Patients noncompliant with therapy, monthly assessed by Pediatric Allergologists, were withdrawn from the study.
  Arms: Oral Viscous Budesonide (OVB)

SUMMARY:
Therapeutic strategies for eosinophilic esophagitis (EoE) actually include: 1) allergen avoidance through dietary modifications, and 2) pharmacologic antiinflammatory therapy. Medical treatment is mainly based on topical administration of corticosteroids by swallowing fluticasone propionate or budesonide spray. Dietetic treatment with highest efficacy is elemental diet, consisting in exclusive feeding with amino-acid based formulas, often administered trough SNG. Alternative choices of acceptable efficacy are empirical six-foods elimination diet (cow's milk, egg, soy, wheat, peanuts, fish) and targeted elimination diet based on the results of allergy tests. Most of the paediatric patients with EE respond to elemental or targeted elimination diets, and therefore such authors recommend elimination diets to be considered the treatment of choice in children. However, elimination diets can often be complex to follow and may be associated with poor adherence owing to the low palatability of a highly restricted diet. In non-compliant patients, especially in adolescents and young adults, it may be more practical to proceed first with corticosteroid treatment. In the case of partial response to elimination diets or corticosteroids, a combination of both treatment mod. However, there has been limited testing of these regimens in randomized controlled trials, while most of available literature is based on case series.

The aim of this study was to compare the efficacy of six-foods elimination diet, swallowed fluticasone, swallowed budesonide and oral viscous budesonide (OVB) in pediatric patients with active EoE. The investigators assessed the effects of randomly assigned treatment on clinical and endoscopic/histologic severity as primary and secondary outcomes, respectively. The investigators describe clinical, allergological, endoscopic and histological features, and pH study results, of our pediatric population.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is characterized by significant eosinophilic infiltration of esophageal mucosa, leading to tissue damage and consequently to esophageal symptoms. The clinical presentation in childhood often mimics gastro-esophageal reflux disease (GERD), sometimes in association to feeding difficulties and failure to thrive. Later in life, the most common symptoms are dysphagia and food impaction, due to esophageal dysmotility. The progression of a non-recognized, untreated disease, is thought to lead to chronic esophageal inflammation with fibrosis and stenosis. Diagnosis requires multiple esophageal biopsies (at least 4 in both proximal and distal esophagus, regardless of gross appearance of mucosa) to demonstrate a mucosal infiltrate of at least 15 eosinophils for high power field (HPF) in patients with a normal pH study or refractory to acid-suppression therapy. Although the endoscopic examination may be unremarkable, endoscopic features of EoE have been well characterized and include: linear furrowing, concentric rings (thachealization), white spots (eosinophilic abscesses), Schatzki ring, strictures, and linear superficial mucosal tears occurring after introduction of the endoscope.

ELIGIBILITY:
Inclusion Criteria:

- suspected, or previously diagnosed, EoE in phase of clinical activity.

Diagnostic criteria were:

1. suggestive esophageal symptoms (GERD-like disease, dysphagia, food impaction);
2. a negative 24 hours pH-impedenzometric study or, whether positive, the refractoriness to a high dose proton pump inhibitor (PPI) therapy for at least 8 weeks;
3. the histological demonstration of >15/20 eosinophils/HPF on at least 1 esophageal biopsy. Patients who received any dietetic or antiinflammatory treatment in the last 6 months were dropped out, and no allergy therapy was allowed during the study

Exclusion Criteria:

* diagnosis of concomitant inflammatory, rheumatic or infectious disease,
* and the assumption of any dietetic or therapy since the clinical onset.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Efficacy Clinical Severity Score | 3 months
  The primary outcome measure was the Clinical Severity Score assessed at baseline (time 0) and after 3 months of treatment (time 1). We scored each symptom basing on its frequency, intensity, and interference on life quality. One point was added in the presence of feeding difficulties leading to growth delay (weight/heigth ratio <5° centile) or significant weight loss (>10% of initial body weight). Two points were added the in case of gastrointestinal bleeding or severe strictures requiring urgent hospitalization.

SECONDARY OUTCOMES:
Efficacy Severity Score for Endoscopy and Histology | 3 months
  Secondary outcome measurements were the Severity Score for Endoscopy and Histology assessed at time 0 and 1

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Pediatrics, Sapienza - University of Rome, Rome, Italy